CLINICAL TRIAL: NCT04108936
Title: Longitudinal Study of the Effect of Cytoreductive Surgery and HIPEC in Patients With Peritoneal Carcinomatoses
Brief Title: Longitudinal Study of CRS/HIPEC for Peritoneal Carcinomatoses
Acronym: CRS/HIPEC
Status: Recruiting | Type: Observational
Sponsor: University of Regensburg (Other)
Collaborators: Krankenhaus Barmherzige Brüder, Regensburg (Other)
Responsible Party: Principal Investigator, Hans J Schlitt, Prof. MD, Head of Surgery, University of Regensburg
Other Study IDs: 15-101-0357
Record Dates: First submitted 2017-02-18; First posted 2019-09-30 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Peritoneal Carcinomatosis
Keywords: CRS; HIPEC; cellular immune response; microbiomes
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples; stool samples; tumor samples; Peritoneal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peritoneal Carcinomatosis: Patients suffering from Peritoneal carcinomatoses from either CRC, gastric cancer or primary peritoneal malignancies
- Control group: Patients suffering from CRC or gastric cancer without peritoneal carcinomatosis

SUMMARY:
Longitudinal Study of the Effect of Cytoreductive Surgery and HIPEC in Patients With Peritoneal Carcinomatoses

DETAILED DESCRIPTION:
Cross-sectional and longitudinal analysis of cellular immune responses in the context of disease outcome.

Cross-sectional and longitudinal analysis of the microbiome in the context of disease outcome.

Analysis of renal function with respect of different HIPEC regimens

Identification of clinical surrogate parameters for outcome.

ELIGIBILITY:
Inclusion Criteria:

* suspicious peritoneal carcinomatosis

Exclusion Criteria:

* <18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicious peritoneal carcinomatosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Through study completion, an average of 3 years
  Prospective analysis of disease free after CRS/HIPEC for peritoneal carcinomatosis
Overall survival | Through study completion, an average of 3 years
  Prospective analysis of overall survival after CRS/HIPEC for peritoneal carcinomatosis

SECONDARY OUTCOMES:
Renal function (serum creatinine (mg/dl)) | Before as well as during the first 7 days postoperative
  Screening for acute renal insufficiency by measuring serum chemistry (serum creatinine (mg/dl) before as well as during the first 7 postoperative days
Renal function (urea (mg/dl)) | Before as well as during the first 7 days postoperative
  Screening for acute renal insufficiency by measuring serum chemistry (serum urea (mg/dl) before as well as during the first 7 days postoperative
Renal function (urine output (ml/24h)) | Before as well as during the first 7 days postoperative
  Screening for acute renal insufficiency by measuring urine output (ml/24h) before as well as during the first 7 postoperative days
Microbiome (Bacterial 16S ribosomal RNA gene sequences will be amplified, sequenced, and analyzed in comparison to publicly available data obtained from healthy volunteers) | Before as well as at postoperative day 2 and 7
  Longitudinal analysis of the microbial burden within samples will be quantified with droplet digital polymerase chain reaction. Bacterial 16S ribosomal RNA gene sequences will be amplified, sequenced, and analyzed in comparison to publicly available data obtained from healthy volunteers.
Cellular immune response (Frequency of NK cell subpopulations within lymphocyte populations measured by flow cytometry) | Before as well as at postoperative day 2 and 7
  Longitudinal analysis of cellular immune responses in blood and peritoneal tissue by flow cytometry. Measuring frequency of NK cell populations within total lymphocyte population
Quality of life (Questionnaire-WHOQOL-BREF) | Before surgery and through study completion, an average of 3 years
  Prospective analysis of quality of life after CRS/HIPEC for peritoneal carcinomatosis. Questionnaire-WHOQOL-BRE produces a quality of life profile. It is possible to derive four domain scores. There are also two items that are examined separately: question 1 asks about an individual's overall perception of quality of life and question 2 asks about an individual's overall perception of their health. The four domain scores denote an individual's perception of quality of life in each particular domain (Physical health (Score 7-35), Psychological (Score 6-30), Social relationships (Score 3-15), Environment (Score 8-40)). Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score transformed to 4-20 or 20-100.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hornung, MD, Study Director — Dept. of Surgery, University Hospital Regensburg; Jens M Werner, MD, Principal Investigator — Dept. of Surgery, University Hospital Regensburg
Locations (2):
- Germany (2):
  - Krankenhaus der Barmherzigen Brüder Regensburg, Regensburg, Bavaria
  - University Hospital Regensburg, Regensburg

REFERENCES:
- [Background] Vivier E, Raulet DH, Moretta A, Caligiuri MA, Zitvogel L, Lanier LL, Yokoyama WM, Ugolini S. Innate or adaptive immunity? The example of natural killer cells. Science. 2011 Jan 7;331(6013):44-9. doi: 10.1126/science.1198687. PMID 21212348
- [Background] Mittal D, Gubin MM, Schreiber RD, Smyth MJ. New insights into cancer immunoediting and its three component phases--elimination, equilibrium and escape. Curr Opin Immunol. 2014 Apr;27:16-25. doi: 10.1016/j.coi.2014.01.004. Epub 2014 Feb 14. PMID 24531241
- [Background] Hoos A, Ibrahim R, Korman A, Abdallah K, Berman D, Shahabi V, Chin K, Canetta R, Humphrey R. Development of ipilimumab: contribution to a new paradigm for cancer immunotherapy. Semin Oncol. 2010 Oct;37(5):533-46. doi: 10.1053/j.seminoncol.2010.09.015. PMID 21074069
- [Background] Sharma P, Wagner K, Wolchok JD, Allison JP. Novel cancer immunotherapy agents with survival benefit: recent successes and next steps. Nat Rev Cancer. 2011 Oct 24;11(11):805-12. doi: 10.1038/nrc3153. PMID 22020206
- [Background] Brahmer JR, Pardoll DM. Immune checkpoint inhibitors: making immunotherapy a reality for the treatment of lung cancer. Cancer Immunol Res. 2013 Aug;1(2):85-91. doi: 10.1158/2326-6066.CIR-13-0078. Epub 2013 Jul 22. PMID 24777499
- [Background] Miller JF, Sadelain M. The journey from discoveries in fundamental immunology to cancer immunotherapy. Cancer Cell. 2015 Apr 13;27(4):439-49. doi: 10.1016/j.ccell.2015.03.007. Epub 2015 Apr 6. PMID 25858803
- [Derived] Kleber J, Yang Zhou J, Weber F, Bitterer F, Hauer P, Kupke P, Kronenberg K, Geissler EK, Schlitt HJ, Hornung M, Hutchinson JA, Werner JM. Immune profile of patients with peritoneal carcinomatosis selected for CRS-HIPEC therapy. Cancer Immunol Immunother. 2023 Nov;72(11):3867-3873. doi: 10.1007/s00262-023-03515-2. Epub 2023 Aug 14. PMID 37580610